CLINICAL TRIAL: NCT05886894
Title: Air Optix Plus HydraGlyde Multifocal Daily/Extended Wear Contact Lenses
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: CLJ241-N003
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Air Optix plus HydraGlyde Multifocal Daily Wear: Lotrafilcon B multifocal soft contact lenses with comfort additive worn in both eyes and removed daily for cleaning and disinfection
  Interventions: Device: Lotrafilcon B multifocal soft contact lenses
- Air Optix plus HydraGlyde Multifocal Extended Wear: Lotrafilcon B multifocal soft contact lenses with comfort additive worn in both eyes worn on an extended wear basis. Extended wear is defined as up to 6 days continuous wear (including while sleeping/overnight).
  Interventions: Device: Lotrafilcon B multifocal soft contact lenses
- Biofinity Multifocal Daily Wear: Comfilcon A multifocal soft contact lenses worn in both eyes and removed daily for cleaning and disinfection
  Interventions: Device: Comfilcon A multifocal soft contact lenses
- Biofinity Multifocal Extended Wear: Comfilcon A multifocal soft contact lenses worn in both eyes worn on an extended wear basis. Extended wear is defined as up to 6 days continuous wear (including while sleeping/overnight).
  Interventions: Device: Comfilcon A multifocal soft contact lenses

INTERVENTIONS:
Device: Lotrafilcon B multifocal soft contact lenses — Commercially available soft (hydrophilic) contact lenses indicated for the correction of presbyopia, with or without myopia or hyperopia
  Other Names: Air Optix plus HydraGlyde Multifocal Daily Wear; Air Optix plus HydraGlyde Multifocal Extended Wear
  Groups: Air Optix plus HydraGlyde Multifocal Daily Wear; Air Optix plus HydraGlyde Multifocal Extended Wear
Device: Comfilcon A multifocal soft contact lenses — Commercially available soft (hydrophilic) contact lenses indicated for the correction of refractive ametropia (myopia and hyperopia) and emmetropia with presbyopia
  Other Names: Biofinity Multifocal Daily Wear; Biofinity Multifocal Extended Wear
  Groups: Biofinity Multifocal Daily Wear; Biofinity Multifocal Extended Wear

SUMMARY:
The purpose of this Post-Market Clinical Follow-Up (PMCF) study is to assess long term performance and safety of Air Optix plus HydraGlyde Multifocal soft contact lenses in a real-world setting when worn as daily wear or extended (overnight) wear.

DETAILED DESCRIPTION:
This is a non-interventional/observational study designed as a retrospective chart review. Study sites will identify charts within their existing databases in a fair and consistent manner, e.g., reviewing all eligible charts in reverse chronological order by year of baseline visit. The baseline visit will be defined as the first office visit where an eye care practitioner provided an in-person office biomicroscopy exam to the patient, before or during which a contact lens prescription for the study or comparator contact lenses was released. Subjects/charts meeting the eligibility criteria will be enrolled in the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Best Corrected Visual Acuity (BCVA) of 20/25 Snellen or better in each eye at baseline;
* Must have worn or be wearing Air Optix plus Hydraglyde Multifocal or Biofinity Multifocal for at least 1 year in a daily wear modality, or 3 years in an extended wear modality;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any recurrent history or active anterior segment infection, inflammation or abnormality contraindicating regular contact lens wear at baseline;
* Use of systemic or ocular medications contraindicating regular contact lens wear at baseline and/or during the period of the retrospective chart collection;
* Slit lamp findings, including signs of pathological dry eye, that would contraindicate regular contact lens wear;
* Participation of the patient in a contact lens or contact lens care product trial during the period of the retrospective chart collection;
* Other protocol-defined exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators will enroll charts following a pre-identified process.
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Distance visual acuity at 1 year - Daily Wear | Year 1
  The subject's chart will be reviewed for distance visual acuity at Year 1, defined as the visit which occurred 1 year (-2/+4 months) since baseline, during which period the subject was wearing the protocol required contact lenses and a contact lens examination was performed. This outcome measure is prespecified for the daily wear arms (Air Optix plus HydraGlyde Multifocal Daily Wear and Biofinity Multifocal Daily Wear).
Near visual acuity at 1 year - Daily Wear | Year 1
  The subject's chart will be reviewed for near visual acuity at Year 1, defined as the visit which occurred 1 year (-2/+4 months) since baseline, during which period the subject was wearing the protocol required contact lenses and a contact lens examination was performed. This outcome measure is prespecified for the daily wear arms (Air Optix plus HydraGlyde Multifocal Daily Wear and Biofinity Multifocal Daily Wear).
Distance visual acuity at 3 years - Extended Wear | Year 3
  The subject's chart will be reviewed for distance visual acuity at Year 3, defined as the visit which occurred 3 years (-2/+8 months) since baseline, during which period the subject was wearing the protocol required contact lenses and a contact lens examination was performed. This outcome measure is prespecified for the extended wear arms (Air Optix plus HydraGlyde Multifocal Extended Wear and Biofinity Multifocal Extended Wear).
Near visual acuity at 3 years - Extended Wear | Year 3
  The subject's chart will be reviewed for near visual acuity at Year 3, defined as the visit which occurred 3 years (-2/+8 months) since baseline, during which period the subject was wearing the protocol required contact lenses and a contact lens examination was performed. This outcome measure is prespecified for the extended wear arms (Air Optix plus HydraGlyde Multifocal Extended Wear and Biofinity Multifocal Extended Wear).
Incidence of corneal infiltrative events - Daily Wear | Up to Year 1
  The subject's chart will be reviewed for incidences of corneal infiltrative events occurring after the baseline exam. This outcome measure is prespecified for the daily wear arms (Air Optix plus HydraGlyde Multifocal Daily Wear and Biofinity Multifocal Daily Wear).
Incidence of corneal infiltrative events - Extended Wear | Up to Year 3
  The subject's chart will be reviewed for incidences of corneal infiltrative events occurring after the baseline exam. This outcome measure is prespecified for the extended wear arms (Air Optix plus HydraGlyde Multifocal Extended Wear and Biofinity Multifocal Extended Wear).
Incidence of microbial keratitis - Daily Wear | Up to Year 1
  The subject's chart will be reviewed for incidences of microbial keratitis occurring after the baseline exam. This outcome measure is prespecified for the daily wear arms (Air Optix plus HydraGlyde Multifocal Daily Wear and Biofinity Multifocal Daily Wear).
Incidence of microbial keratitis - Extended Wear | Up to Year 3
  The subject's chart will be reviewed for incidences of microbial keratitis occurring after the baseline exam. This outcome measure is prespecified for the extended wear arms (Air Optix plus HydraGlyde Multifocal Extended Wear and Biofinity Multifocal Extended Wear).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (8):
- United States (8):
  - Complete Family Vision Care, San Diego, California
  - Pearle Vision, Jacksonville, Florida
  - Jackson Health Community Center, Miami, Florida
  - Vision Health Institute, Orlando, Florida
  - Complete Eye Care of Medina, Medina, Minnesota
  - Koetting Associates, St Louis, Missouri
  - Sacco Eye Group, Vestal, New York
  - Smith Bowman Ophthalmology, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No